CLINICAL TRIAL: NCT05508802
Title: Interventional Cooperative Agreement Program - Vocational Intervention Demonstration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: L-1171-21B
Record Dates: First submitted 2022-01-19; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries; Brain Injuries; Employment; Spinal Cord Diseases
Keywords: employment; vocational rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries; Spinal Cord Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- State Counselor-Coordinated Services (Other): In this program, services are coordinated by a counselor employed by the New Jersey State Division of Vocational Rehabilitation Services (NJDVRS), a state-based agency that assists people with disabilities who are interested in pursuing employment. While the participant is in inpatient rehabilitation or soon after their discharge, a member of the research team will assist them in completing the necessary documentation to apply for services from this agency. Services for which they are eligible will be provided directly through NJDVRS.
  Interventions: Other: State Counselor-Coordinated Services
- Center Facilitator-Coordinated Services (Other): In this program, services are coordinated by a facilitator who is employed by Kessler Institute for Rehabilitation and works cooperatively with NJDVRS. The facilitator will begin working with the participant during inpatient rehabilitation, or soon after discharge, depending on when they enroll in the study. Some services for which they are eligible will be provided through NJDVRS and others will be provided to them by the facilitator.
  Interventions: Other: Center Facilitator-Coordinated Services

INTERVENTIONS:
Other: State Counselor-Coordinated Services — A counselor affiliated with the New Jersey State Division of Vocational Rehabilitation Services coordinates services that consider the participant's condition, needs and goals. Services they may receive include:
  * Education on programs designed to help people with spinal cord injury or brain injury pursue employment.
  * Advice and guidance from professional counselors who have special training in helping people with disabilities pursue employment.
  * Help completing applications for services.
  * Assistance communicating with my employer about my needs and ways to accommodate them.
  * Referrals to and services from other health care or technology providers.
  Arms: State Counselor-Coordinated Services
Other: Center Facilitator-Coordinated Services — A facilitator affiliated with Kessler Institute for Rehabilitation coordinates services that consider the participant's condition, needs and goals. Services they may receive include:
  * Education on programs designed to help people with spinal cord injury or brain injury pursue employment.
  * Advice and guidance from professional counselors who have special training in helping people with disabilities pursue employment.
  * Help completing applications for services.
  * Assistance communicating with my employer about my needs and ways to accommodate them.
  * Referrals to and services from other health care or technology providers.
  Arms: Center Facilitator-Coordinated Services

SUMMARY:
For many people with spinal cord injury or brain injury, seeking employment after injury is an important goal. There are services available to help people with disabilities. However, the best ways to coordinate and deliver these services are not yet known. This project will compare two ways of coordinating and delivering services that are designed to help people with spinal cord injury or brain injury obtain employment.

DETAILED DESCRIPTION:
Employment is important for financial security, social connection, and life satisfaction. Unfortunately, rates of unemployment remain high among people with spinal cord injury (SCI) and brain injury (BI). To help address this challenge, the investigators are conducting a single-site, randomized, controlled trial to compare two programs intended to increase rates of employment among people with SCI or BI. In one program, services are coordinated by a counselor employed by the New Jersey State Division of Vocational Rehabilitation Services, a state-based agency that assists people with disabilities who are interested in pursuing employment. In the other program, services are coordinated by a facilitator who is employed by the rehabilitation hospital at which the participant receives inpatient care. Services provided in both programs will be customized to the participant's needs and goals. Services will begin in inpatient rehabilitation and may include education, therapy, equipment provision, counseling, and other interventions.

The project will enroll 500 participants who are interested in becoming employed or returning to work. Information about employment status, earnings, benefits use, community participation, and health will be collected through a combination of surveys, medical record review, and information available in state and federal administrative databases. Analyses will examine the rate of participants employed at 1 year after enrollment in each group, time to employment, earnings, benefits usage, community participation, and well-being. Findings from this study will be used to determine which ways of delivering services are most effective in enabling employment, and to provide information to help other rehabilitation centers adopt effective programs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-62
* New Jersey resident
* Admitted to Kessler Institute for Rehabilitation (KIR) due to a spinal cord injury (SCI) or brain injury (BI)
* Receiving inpatient rehabilitation at KIR
* Community living in the state of New Jersey after discharge from KIR

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Employment Status | 12-months post-enrollment
  Proportion of participants in each group in competitive employment

SECONDARY OUTCOMES:
Earnings | 12-months post-enrollment
  Earnings within the first 12 months post-enrollment as obtained from New Jersey Unemployment Insurance (UI) data
SSI and SSDI Benefit Applications | 12-months post-enrollment
  Proportion of participants who report via survey that they applied for Supplemental Security Income (SSI) and Social Security Disability Insurance (SSDI) benefits
SSI and SSDI Benefit Awards | 12-months post-enrollment
  Proportion of participants who report via survey that they were awarded SSI and SSDI benefits
Job Satisfaction | 12-months post-enrollment
  Survey to assess job satisfaction and attitudes toward work
Satisfaction with Services | 12-months post-enrollment
  Survey to assess satisfaction with services provided
Self-Reported Health and Well-Being | 12-months post-enrollment
  Survey to assess emotional well-being, current general health status, and extent to which current health limits ability to work

IPD SHARING:
Plan to Share IPD: No